CLINICAL TRIAL: NCT00529321
Title: Open-label, Dose-escalating, Phase I Study of TG4040 (MVA-HCV) in Treatment-naïve Patients Chronically Infected With Hepatitis C Virus (HCV Genotype 1)
Brief Title: Immunotherapy With TG4040 in Treatment-naïve Patients Chronically Infected With Hepatitis C Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Transgene (Industry)
Responsible Party: Transgene, Transgene
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG4040.01
Record Dates: First submitted 2007-09-07; First posted 2007-09-14 (Estimated); Last update posted 2010-09-03 (Estimated); Status verified 2010-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Immunotherapy

INTERVENTIONS:
Biological: MVA-HCV (Immunotherapy) — MVA-HCV

SUMMARY:
The primary objective is to determine the safety of sub-cutaneous (SC) injections of TG4040 in non-cirrhotic, treatment-naïve patients chronically infected with HCV (genotype 1).

Patients will be sequentially treated at an escalting dose of TG4040. All patients will be followed up to at least 6 months after his/her first injection. In addition, all patients treated at the highest dose will receive a TG4040 boost injection 6 months after the first injection, and will be followed up during an additional 6-month period.

DETAILED DESCRIPTION:
The first nine patients will be sequentially treated in three cohorts of three patients, i.e. they will receive 3 SC injections of TG4040 on Days 1, 8 and 15, at the dose of 10e6 pfu (first cohort), 10e7 pfu (second cohort), or 10e8 pfu (third cohort).

There will be a one-week safety interval between the first injection of the patients of a given cohort, and a two-week safety interval between the last injection of the last patient of a given cohort and the first injection of the first patient of the next one. There will be also a two-week safety observation period after the last injection of the last patient of the third cohort. If the dose of 10e8 pfu does not raise safety problems, then 6 patients will be further enrolled, without safety intervals between patients. They will receive 3 SC injections of TG4040 at the dose of 10e8 pfu, on Days 1, 8 and 15.

All patients will be followed up to at least 6 months after his/her first injection. In addition, all patients treated at the dose of 10e8 pfu will receive a TG4040 boost injection 6 months after the first injection, and will be followed up during an additional 6-month period.

Three additional cohorts of 9 patients will receive a boost injection either at 2, 4 or 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained and signed;
* Male or female patients;
* With chronic hepatitis C (genotype 1) evidenced by HCV positive serology detectable for more than 6 months;
* Patients with fibrosis status graded F0 or F1 according to the METAVIR grading system; patients with a F2 fibrosis stage could be enrolled on a case-by-case basis after being sure that they have a contraindication to be treated with an IFN-based standard HCV treatment; patients with F3 or F4 fibrosis stage will not be enrolled; this will be assessed either on the liver biopsy performed less than 18 months prior to baseline or on a FibroTest® and a FibroScan® performed within 2 months prior to first TG4040 injection; in case of discordant results, a liver biopsy will be performed prior to TG4040 treatment;;
* Treatment-naïve patients: patients who have never received IFN-based treatment;
* Patients must have compensated liver disease, with:

  * No history of ascites, hepatic encephalopathy or bleeding from esophageal varices;
  * Laboratory tests values:

    * Serum alanine aminotransferase (ALT)less then 2 folds the Upper Limit of Normal (ULN);
    * Serum bilirubin and international normalized ratio (INR) values within normal range (except in patients with Gilbert syndrome where serum bilirubin may be as high as 3.0 mg/dL); and
    * Other laboratory parameters of grade 0 or 1 (CTC criteria);
* For women of child-bearing potential, i.e. with no history of hysterectomy or tubal ligation, a negative pregnancy test at study entry and adequate protection against pregnancy during the conduct of the study and until 3 months after last TG4040 injection.

Additionnal cohorts:

* Patients with high ALT level (2 folds ULN<ALT<5 folds ULN in the 2 months before inclusion) and fibrosis not higher than F2.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* Co-infection with HBV (indicated by the presence of Hepatitis B Surface Antigen (HBsAg) in serum; patients with anti-hepatitis B core antibody response (anti-HBc) will not be excluded) or HIV (anti-HIV antibodies in serum); patients with HIV positive sexual partner (by history) will not be included;
* Current HCV therapies;
* Active IV drug or alcohol abuse;
* Serious, concomitant disorder, including:

  * primary biliary cirrhosis or sclerosing cholangitis;
  * auto-immune disease such as symptomatic cryoglobulinemia, polyarthritis, multiple sclerosis; a broad auto-immune testing will be performed at baseline;
  * proven or suspected immunosuppressive disorder;
  * active systemic infection; if the patient has acute febrile illness ( > 38°C) on the day of vaccination, it will be delayed by at least one week after complete recovery;
* Malignancy within the last 5 years; patients with history of squamous cell skin cancer or basal cell skin cancer will be enrolled, unless the history of skin cancer is at the vaccination site;
* Systemic corticosteroid therapy or other immunosuppressive/immunomodulating drugs (e.g. Cyclosporine) within 2 months prior to first study drug injection; corticosteroid nasal sprays, inhaled steroids for asthma and/or topical steroids are permissible;
* Participation in another experimental protocol during the study period (last intake of investigational drug within 6 months prior to baseline);
* Breast-feeding women;
* Receipt of any inactivated vaccine 14 days prior to vaccination or for the duration of the study; receipt of any live attenuated vaccine within 30 days prior to vaccination or for the duration of the study;
* Allergy to eggs;
* Patient unable to comply with the protocol requirements;
* Any condition that, in the opinion of the investigator, might interfere with study objectives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events, vital signs, physical examination, standard laboratory tests) | regularly

SECONDARY OUTCOMES:
Virology (quantification of HCV-RNA), immunology (cellular-mediated and humoral immune responses) | regularly

CONTACTS AND LOCATIONS:
Overall Officials: Christian TREPO, MD, Principal Investigator — Hopital de l'Hotel-Dieu
Locations (6):
- France (6):
  - Hôpital Henri Mondor, Créteil
  - Hopital A. Michallon, La Tronche
  - Hopital de l'Hotel-Dieu, Lyon
  - Hôpital de l'Hôtel Dieu, Nantes
  - Hopital Civil, Strasbourg
  - Hôpital de Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Habersetzer F, Honnet G, Bain C, Maynard-Muet M, Leroy V, Zarski JP, Feray C, Baumert TF, Bronowicki JP, Doffoel M, Trepo C, Agathon D, Toh ML, Baudin M, Bonnefoy JY, Limacher JM, Inchauspe G. A poxvirus vaccine is safe, induces T-cell responses, and decreases viral load in patients with chronic hepatitis C. Gastroenterology. 2011 Sep;141(3):890-899.e1-4. doi: 10.1053/j.gastro.2011.06.009. Epub 2011 Jun 13. PMID 21699798
- See also: Related Info — http://www.nlm.nih.gov/medlineplus/hepatitisc.html